CLINICAL TRIAL: NCT07025044
Title: Characterizing the Postmenopausal Genitourinary Microbiome in Women Undergoing Onabotulinum Toxin Type A for Overactive Bladder - A Feasibility Trial
Brief Title: Assessing the Genitourinary Microbiome of Women With Overactive Bladder Undergoing Onabotulinum Toxin Type A Intradetrusor Injections
Acronym: MICROAB_Pilot
Status: Recruiting | Type: Observational
Sponsor: Alexis Dieter (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor-Investigator, Alexis Dieter, Attending Physician, MedStar Health
Organization: Medstar Health Research Institute (Other)
Other Study IDs: STUDY00009131
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder (OAB); Urge Incontinence
Keywords: onabotulinum toxin type A
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women >55yo undergoing onabotulinum toxin type A injection for OAB in clinic
  Interventions: Drug: onabotulinum toxin type a

INTERVENTIONS:
Drug: onabotulinum toxin type a — All subjects will be scheduled to undergo Onabotulinum toxin type A intradetrusor injection for management of OAB. On Day 0, subjects will undergo Onabotulinum toxin type A injection by a licensed clinical provider and receive a one-time dose of Nitrofurantoin for infection prevention per standard clinic protocol.
  Other Names: Botox; BTX

SUMMARY:
Single-site prospective observational pilot feasibility study of women with overactive bladder/urge urinary incontinence undergoing onabotulinum toxin type A intradetrusor injections in order to achieve the following objectives:

* Establish a record of successful collaboration with Dr. Ravel, an expert researcher in the female microbiome based at the University of Maryland
* Demonstrate the investigators' ability to recruit subjects from the diverse population of postmenopausal women undergoing BTX for OAB within MedStar Health Urogynecology clinics
* Collect, process and analyze urine specimens collected prior to and 4-weeks after BTX injection, and to compare the GU microbiome of self-collected versus clinic-collected samples
* Assess response to BTX treatment and explore rates of and risk factors for urinary tract infection and incomplete voiding requiring catheterization within the first 4-weeks after BTX

DETAILED DESCRIPTION:
Participants will be recruited from MedStar Urogynecology clinics. English-speaking postmenopausal natal female > 55 years old scheduled to undergo BTX for treatment of overactive bladder (OAB) will be eligible for enrollment.

All subjects will be scheduled to undergo Onabotulinum toxin type A intradetrusor injection for management of OAB. On Day 0, subjects will undergo BTX injection by a licensed clinical provider and receive a one-time dose of Nitrofurantoin for infection prevention per standard clinic protocol. Per standard clinic protocol, all patients undergoing BTX receive a one-time dose of oral nitrofurantoin for infection prevention unless they have allergy/contraindication to nitrofurantoin or they are at high risk of UTI (3 or more culture-proven UTIs in the past year). BTX dose, any prior BTX treatments and time since last BTX injection will be recorded.

Voided urine specimens will be collected at the baseline and follow-up visits. Each subject will be asked to complete one self-collection and one clinic-collection at each time point for a total of four collections over the course of the study

Sample size is 40 subjects in this pilot feasibility study. Subjects will be followed for approximately 1 month after BTX injection. Self-collected and clinic-collected urine specimens will be obtained at baseline and 4 weeks after BTX injection. Subjects will also complete baseline questionnaires and validated patient reported outcome measures at baseline and 4 weeks follow-up. Subjects will be provided reimbursement for parking costs ($17/visit) for the procedure visit and for the follow-up visit. Subjects will be provided a payment of $50 upon completion of the follow-up visit activities.

ELIGIBILITY:
Inclusion Criteria:

* Natal female > 55 years old
* English-speaking
* Scheduled to undergo onabotulinum toxin type A for treatment of OAB
* No menses for >1 year if uterus in situ
* Planning one dose nitrofurantoin for antibiotic prophylaxis at time of onabotulinum toxin type A injection per clinic protocol

Exclusion Criteria:

* Diagnosis of painful bladder syndrome
* Current symptomatic or clinically-suspected UTI within 30 days prior to onabotulinum toxin type A injection procedure*
* Systemic antibiotic exposure within 30 days^
* Prophylactic antibiotic treatment for recurrent UTI within the last 12 months
* Current systemic immunosuppressive therapy (i.e. prednisone or immunomodulators) immunotherapy, chemotherapy or radiation treatment
* Prior pelvic radiation
* Indwelling catheter or intermittent catheterization

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from the patient population treated at a MedStar Urogynecology clinics located across DC, Maryland and Virginia will be recruited and eligible for enrollment. Potential subjects will be identified both via provider referral and through electronic medical record review to identify patients scheduled for onabotulinum toxin type A injection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 6 months
  recruitment of 40 eligible subjects from our diverse population of postmenopausal women undergoing BTX for OAB

SECONDARY OUTCOMES:
Urine sample collection and comparison | 4 weeks
  To collect, process and analyze urine specimens collected prior to and 4-weeks after BTX injection, and to compare the GU microbiome of self-collected versus clinic-collected samples
Onabotulinum toxin type A response | 4 weeks
  To assess response to Onabotulinum toxin type A treatment 4-weeks after Onabotulinum toxin type A
Onabotulinum toxin type A adverse events | 4 weeks
  To explore rates of and risk factors for UTI and incomplete voiding requiring catheterization within the first 4-weeks after Onabotulinum toxin type A injection

OTHER OUTCOMES:
International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) score | 4 weeks
  Validated questionnaire score used to evaluate female lower urinary tract symptoms and impact on quality of life using the International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (ICIQ-FLUTS), a 12-item questionnaire used to evaluate female lower urinary tract symptoms and impact on quality of life. The ICIQ-FLUTS asks respondents to rate the frequency of a specific lower urinary tract symptom (such as urgency, frequency, pain, etc.) on various five-point scales and then asks the subject to rate the level of bother from that specific symptom on a Likert scale from (0) "not at all" to (10) "a great deal." Higher score = more bother.
Pelvic Floor Distress Inventory-20 (PFDI-20) score | 4 weeks
  20-item condition-specific quality-of-life instrument with three scales (6-item Urinary Distress Inventory, 6-item Pelvic Organ Prolapse Distress Inventory, and 8-item Colorectal-Anal Distress Inventory) used to evaluate the impact of pelvic floor disorders on quality of life. The UDI-6 is a preferred PRO for assessing female UI. A higher score = more distress. The patient acceptable symptom state (PASS) for the UDI-6 is < 37.5.
Incontinence Impact Questionnaire Short Form (IIQ-7) score | 4 weeks
  7-item condition-specific quality-of-life instrument assessing impact of urinary symptoms on quality of life. Higher score = more impact (worse symptoms). The PASS threshold for the IIQ-7 is < 33.3
Patient Global Impression of Severity (PGI-S) | 4 weeks
  A single item questionnaire to assess a person's impression of disease severity. Higher score = more severe disease. The PASS threshold for the PGI-S is < 3.
Accountable Health Communities Health-Related Social Needs Screening Tool (AHC HRSN) | Baseline
  10-item screening tool designed by the Centers for Medicare & Medicaid Services Center for Medicare and Medicaid Innovation to assess health-related social needs across five core domains - housing instability, food insecurity, transportation problems, utility help needs, and interpersonal safety. Higher score = worse score.
Patient Global Impression of Improvement (PGI-I) | 4 weeks
  a single item questionnaire to assess an individual's impression of change in urinary symptoms on a 7-point Likert scale ranging from (1) "very much better" to (7) "very much worse." The PASS threshold for the PGI-I is < 3. Lower score = more improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Urogynecology Clinic, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No